CLINICAL TRIAL: NCT04999267
Title: A Tailored School-based Intervention to INcrease VaccinE Uptake Among adoleScenTs (INVEST) in the Rural South
Brief Title: Increasing Vaccine Uptake Among Adolescents in the Rural South
Acronym: INVEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00101137
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Vaccine Hesitancy
Keywords: Human papillomavirus (HPV); Adolescent; School based intervention; Vaccine; HPV vaccine
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INVEST Intervention School Districts (Experimental)
  Interventions: Other: INVEST

INTERVENTIONS:
Other: INVEST — The intervention will consist of 3 primary components: 1) school nurse training and technical support for promoting adolescent vaccination (Tdap, MenACWY, HPV) and strengthening existing school nursing vaccination programming, 2) caregiver-targeted educational materials that are disseminated via school nurses, and 3) tools and resources to facilitate linkage to vaccination providers in the local community. Existing materials will be used in the intervention such as resources available from the Centers for Disease Control and Prevention and Middle School Health Starts Here tool kit from the National Association of School Nurses and the National HPV Roundtable. Technical support includes the study team working with local school nurses to identify educational materials available from national and statewide sources.

SUMMARY:
The benefits of adolescent vaccines are well known for preventing meningococcal infection and human papillomavirus (HPV)-related pre-cancerous lesions. Yet, many adolescents in the United States (US) remain under-vaccinated, with vaccination rates among rural adolescents significantly lower than among their urban peers. In addition, there are urban-rural disparities in the coverage of HPV vaccine, particularly in Southern states like North and South Carolina, which currently fall below the Healthy People 2020 goal of ≥80% coverage. The goal of the proposed study is to evaluate the feasibility and preliminary efficacy of a school-based intervention for increasing vaccine uptake among adolescents in rural North and South Carolina.

ELIGIBILITY:
Inclusion Criteria:

- Any public middle school in Cherokee County, South Carolina or Rockingham County, North Carolina school districts

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Walter, MD, MPH, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - University of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: School nurses from intervention schools were not considered enrolled.
Units Other Than Participants: School District
Period: Overall Study
Arm/Group | INVEST Intervention School Districts
Started | 2868; 2 School District
Completed | 2868; 2 School District
Not Completed | 0; 0 School District

BASELINE CHARACTERISTICS:
Population: The participants are school districts; baseline characteristics data were not collected.
Groups:
- INVEST Intervention: INVEST: The intervention will consist of 3 primary components: 1) school nurse training and technical support for promoting adolescent vaccination (Tdap, MenACWY, HPV) and strengthening existing school nursing vaccination programming, 2) caregiver-targeted educational materials that are disseminated via school nurses, and 3) tools and resources to facilitate linkage to vaccination providers in the local community. Existing materials will be used in the intervention such as resources available from the Centers for Disease Control and Prevention and Middle School Health Starts Here tool kit from the National Association of School Nurses and the National HPV Roundtable. Technical support includes the study team working with local school nurses to identify educational materials available from national and statewide sources.
Arm/Group | INVEST Intervention
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Percentage of Adolescents Who Ever Received at Least One Dose of HPV Vaccination in the Intervention Group After the Intervention Implementation Compared With Before Intervention Implementation
Description: HPV vaccination status (received at least one versus no doses) of middle schoolers (by district) will be obtained from official vaccination records before and after intervention implementation.
Time Frame: Baseline, 9 months
Measure: Number; unit: percentage of adolescents
Units Other Than Participants: School District
Arm/Group | INVEST Intervention
Number analyzed (Participants) | 2868
Number analyzed (School District) | 2
percentage of adolescents | 21.7
Statistical Analysis 1: Comparison: INVEST Intervention; Test type: Other — Pre-intervention vs. Post-intervention analysis; p < 0.0001, Chi-squared

2. Secondary Outcome: Difference in Percentage of Adolescents Who Have Completed the HPV Vaccination Series (2 Doses Depending on Age at Vaccination Initiation) in the Intervention Group After Implementation Compared With Before Intervention Implementation
Description: as for outcome 1
Time Frame: Baseline, 9 months
Measure: Number; unit: percentage of adolescents
Units Other Than Participants: School District
Arm/Group | INVEST Intervention
Number analyzed (Participants) | 2868
Number analyzed (School District) | 2
percentage of adolescents | 7.6
Statistical Analysis 1: Comparison: INVEST Intervention; Test type: Other — Pre-intervention vs. Post-intervention analysis; p < .0001, Chi-squared

3. Secondary Outcome: Fidelity of Intervention Across Intervention Schools
Description: Score items (0-100%) from a study specific checklist (Fidelity Checklist) will be completed by school nurses from intervention schools with a high score (100%) indicating more adherence to the study intervention and 0% indicating the worse score and less adherence to the study intervention
Time Frame: 9 months
Population: School nurses from intervention schools.
Measure: Mean (Full Range); unit: Percent
Units Other Than Participants: School District
Arm/Group | INVEST Intervention
Number analyzed (Participants) | 88
Number analyzed (School District) | 2
Percent | 87.5 [76.1 to 98.9]

ADVERSE EVENTS:
Time Frame: Participants are school districts, therefore no adverse events were collected.
Description: Participants are school districts, therefore no adverse events were collected.
Arm/Group | INVEST Intervention
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04999267/Prot_SAP_002.pdf
  • Informed Consent Form (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT04999267/ICF_000.pdf